CLINICAL TRIAL: NCT00966225
Title: An Open-label Dose-finding Study of LIP-01 in Otherwise Healthy Individuals With Hypercholesterolemia
Brief Title: LIP-01 in Hypercholesterolemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Afexa Life Sciences Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LIP-01-2009-1
Record Dates: First submitted 2009-08-18; First posted 2009-08-26 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- One gram LIP-01 per day (Experimental): One gram LIP-01 per day for 12 weeks
  Interventions: Dietary Supplement: LIP-01
- Two grams LIP-01 per day (Experimental): Two grams LIP-01 per day for 12 weeks
  Interventions: Dietary Supplement: LIP-01
- 0.333 grams LIP-01 per day (Experimental): 0.333 grams LIP-01 per day for 12 weeks
  Interventions: Dietary Supplement: LIP-01

INTERVENTIONS:
Dietary Supplement: LIP-01 — comparison of different dosages of natural health product

SUMMARY:
The purpose of this study is to determine a safe and tolerable dose of LIP-01

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-75 years
* Plasma total-cholesterol >5.2 mmol/L (> 200 mg/dL)
* Willingness to adhere to the requirements of the protocol, including availability for follow-up visits and donation of blood samples
* Willingness and ability to sign written informed consent
* Women of child bearing capacity who agree to use an acceptable form of birth control during the trial [i.e., oral contraception, reliable use of a double-barrier method (e.g., condom and diaphragm, condom and foam, condom and sponge), IUD or tubal ligation]

Exclusion Criteria:

* Plasma triglycerides > 4.0 mmol/L (> 354 mg/dL)
* Plasma LDL ≥ 5.0 mmol/L (≥ 195 mg/dL)
* Current coronary artery/ cardiovascular disease or history of a cardiovascular event (stroke, transient ischemic attack, myocardial infarction, angioplasty or coronary artery bypass grafting, angina pectoris)
* Moderate/high risk of coronary artery/ cardiovascular disease
* Diabetes mellitus
* Uncorrected hypothyroidism
* Other significant metabolic endocrine disease
* Uncontrolled hypertension (>160 systolic or >100 diastolic)
* Active liver disease (ALT >2x normal)
* Significant gastrointestinal disease
* Acute inflammatory disease
* Significant kidney disease (calculated by eGFR <60 mL/min)
* Any other significant medical condition which, in the opinion of the investigator, could compromise patient safety or confound trial results
* Any significant/relevant surgery within the last year
* Use of lipid-lowering drugs
* Treatment within the previous 6 months with any medication that is known to affect lipid or lipoprotein levels (such as statins, fibric acid derivatives, bile acid sequestrants, ezetimibe, nicotinic acid)
* Regular use of natural health products or dietary supplements known to affect lipid or lipoprotein levels (omega-3 fatty acids, green tea extracts, guggulipid, psyllium, plant sterols, policosanols). If the participants agree to stop taking these products prior to study entry and for the duration of the study, they can participate in the study.
* Pregnant or lactating women
* Known allergy to any ingredient in the study product, including: Coptis chinensis, Ilex kudingcha, microcrystalline cellulose and magnesium stearate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
To determine a safe and tolerable dose of LIP-01 | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lewanczuk, MD, PhD, FRCPC, Principal Investigator — University of Alberta
Locations (2):
- Medicus Research, LLC, Northridge, California, United States
- The Northern Alberta Clinical Trials and Research Centre, Edmonton, Alberta, Canada